CLINICAL TRIAL: NCT01482221
Title: A Multicenter, Randomized, Double-blind, Parallel Group, Placebo-controlled, Phase IIb Efficacy and Safety Study of Adjunctive AZD6765 in Patients With Major Depressive Disorder (MDD) and a History of Inadequate Response to Antidepressants
Brief Title: A Study to Assess the Effect and Safety of AZD6765 in Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D6702C00031; EudraCT number 2011-004690-87
Record Dates: First submitted 2011-11-28; First posted 2011-11-30 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; MDD; Inadequate Response to Antidepressant Therapy; Channel blocker of the NMDA class of glutamate receptors
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: AZD6765 iv
- 2 (Experimental)
  Interventions: Drug: AZD6765 iv
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD6765 iv — 50 mg (AZD6765 Solution for Infusion, 0.5 mg/mL) by iv infusion.
  Arms: 1
Drug: AZD6765 iv — 100 mg (AZD6765 Solution for Infusion, 1.0 mg/mL) by iv infusion.
  Arms: 2
Drug: Placebo — 0.9 sodium chloride [normal saline] solution for injection by iv infusion
  Arms: 3

SUMMARY:
The purpose of this study is to assess the effect and safety of AZD6765 in patients with major depressive disorder who exhibit inadequate response to antidepressants. AZD6765 is a channel blocker of the N-methyl-D-aspartate (NMDA) class of glutamate receptors.

DETAILED DESCRIPTION:
A Multicenter, Randomized, Double-blind, Parallel Group, Placebo-controlled, Phase IIb Efficacy and Safety Study of Adjunctive AZD6765 in Patients with Major Depressive Disorder (MDD) and a History of Inadequate Response to Antidepressants

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent before initiation of any study-related procedures.
* Male or female patients aged 18 to 70 years, inclusive.
* The patient must have a clinical diagnosis of major depressive disorder with a lifetime history of inadequate response to at least 3 antidepressants.
* Women of child-bearing potential must have a negative serum pregnancy test and confirmed use of a highly effective form of birth control before enrollment for a minimum of 3 months before study start.
* Outpatient status at screening and randomization visits.

Exclusion Criteria:

* Patients with a history of diagnosed bipolar disorder or schizophrenia or schizoaffective disorder or currently exhibiting psychotic features associated with their depression; dementia or suspicion thereof.
* Patients who have had a suicide attempt within the last 6 months.
* Electroconvulsive therapy (ECT), vagal nerve stimulation (VNS) or transcranial magnetic stimulation (TMS) or previous treatment with ketamine infusion within the 6 months prior to screening, or any history of deep brain stimulation.
* Patients with any history of seizure disorder (except for febrile seizures in childhood).
* Pregnancy or lactation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 542 (Actual)
Dates: Start 2011-12-16 (Actual); Primary Completion 2013-08-26 (Actual); Study Completion 2013-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dhaval A Desai, MD, Study Director — 1800 Concord Pike, Wilmington, DE 19850
Locations (44):
- United States (33):
  - Research Site, Chino, California
  - Research Site, Lond Beach, California
  - Research Site, San Diego, California
  - Research Site, Stanford, California
  - Research Site, New Heaven, Connecticut
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Gainsville, Florida
  - Research Site, Lake City, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Decatur, Georgia
  - Research Site, Hoffman Estates, Illinois
  - Research Site, Joliet, Illinois
  - Research Site, Skokie, Illinois
  - Research Site, Lake Charles, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Minneapolis, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Willingboro, New Jersey
  - Research Site, Mount Kisco, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Bellevue, Washington
- Chile (2):
  - Research Site, Antofagasta
  - Research Site, Santiago
- Slovakia (6):
  - Research Site, Bratislava
  - Research Site, Liptovský Mikuláš
  - Research Site, Michalovce Stranany
  - Research Site, Rimavská Sobota
  - Research Site, Svidník
  - Research Site, Trnava
- South Africa (3):
  - Research Site, Cape Town
  - Research Site, Johannesburg
  - Research Site, Tygervalley

REFERENCES:
- See also: D6702C00031_Clinical Study Report_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=575&filename=D6702C00031_AZD6765_CSR_Synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study was conducted in Chile, Slovakia, South Africa, and the United States between 16 December 2011 and 26 August 2013. A total of 542 patients were enrolled in the study and of these, 302 patients were randomized to treatment. 240 patients were not randomized to treatment due to eligibility criteria not being fulfilled.
Pre-assignment Details: The study had a screening/washout period of up to 42 days, a 12-week double blind treatment period, and a 14-day follow-up period. Patients received 3 infusions per week during Weeks 1 to 3,1 infusion per week during Weeks 4 to 6, and 1 infusion every other week during Weeks 7 to 12.
Groups:
- AZD6765 50 mg; AZD6765 100 mg; Placebo: Intravenous infusion
Period: Overall Study
Arm/Group | AZD6765 50 mg | AZD6765 100 mg | Placebo
Started | 101 | 101 | 100
Completed | 80 | 81 | 77
Not Completed | 21 | 20 | 23
Not completed — Lack of Efficacy | 1 | 0 | 1
Not completed — Lost to Follow-up | 3 | 2 | 1
Not completed — Study-Specific Withdrawal Criteria | 2 | 0 | 1
Not completed — Condition under Investigation Worsened | 3 | 2 | 4
Not completed — Severe Non-Compliance to Protocol | 1 | 0 | 1
Not completed — Adverse Event | 1 | 7 | 3
Not completed — Withdrawal by Subject | 10 | 7 | 12
Not completed — Incorrect randomization | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD6765 50 mg | AZD6765 100 mg | Placebo | Total
Number analyzed (Participants) | 101 | 101 | 100 | 302
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.7 (11.19) | 47.5 (11.89) | 49.5 (11.12) | 48.2 (11.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 70 | 65 | 197
  Male | 39 | 31 | 35 | 105
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 91 | 87 | 91 | 269
  Black or African American | 8 | 11 | 6 | 25
  Asian | 0 | 3 | 1 | 4
  Other | 2 | 0 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 6 in the Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: A 10-item scale for the evaluation of depressive symptoms. Each MADRS item is rated on a 0 to 6 scale. The MADRS total score is calculated as the sum of the 10 individual item scores; the total score can range from 0 to 60. Higher MADRS scores indicate higher levels of depressive symptoms.
Time Frame: Baseline to Week 6
Population: The modified intent-to-treat (mITT) analysis set included all randomized patients, who took investigational product (IP) and who have a non-missing baseline MADRS total score and at least 1 post-baseline MADRS total score, classified according to their randomized treatment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | AZD6765 50 mg | AZD6765 100 mg | Placebo
Number analyzed (Participants) | 101 | 100 | 97
units on a scale | -14.37 (1.238) | -14.40 (1.244) | -13.18 (1.266)
Statistical Analysis 1: Comparison: AZD6765 50 mg vs Placebo; Mixed model repeated measures (MMRM) includes treatment, pooled center, visit, treatment by visit interaction, and baseline MADRS score by visit interaction as explanatory variables. Treatment, visit, treatment by visit interaction, and baseline MADRS score by visit interaction are fixed effects in the model; pooled center is a random effect; Test type: Superiority or Other; p = 0.630, Mixed models for repeated measures — The adjusted p-values protect the overall family-wise error rate across the 6 key comparisons of AZD6765 100 mg and 50 mg to placebo (for MADRS change from baseline to 6 weeks and to 12 weeks and for Sustained Response); LS mean difference = -1.18, 95% CI 2-sided [-4.519 to 2.152], Standard Error of Mean 1.695
Statistical Analysis 2: Comparison: AZD6765 100 mg vs Placebo; MMRM includes treatment, pooled center, visit, treatment by visit interaction, and baseline MADRS score by visit interaction as explanatory variables. Treatment, visit, treatment by visit interaction, and baseline MADRS score by visit interaction are fixed effects in the model; pooled center is a random effect; Test type: Superiority or Other; p = 0.476, Mixed models for repeated measures — [p-value comment as in outcome 1, analysis 1]; LS mean difference = -1.21, 95% CI 2-sided [-4.563 to 2.134], Standard Error of Mean 1.701

2. Secondary Outcome: Change From Baseline to Week 12 in the Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: as for outcome 1
Time Frame: Baseline to Week 12
Population: The modified intent-to-treat (mITT) analysis set included all randomized patients, who took IP and who have a non-missing baseline MADRS total score and at least 1 post-baseline MADRS total score, classified according to their randomized treatment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | AZD6765 50 mg | AZD6765 100 mg | Placebo
Number analyzed (Participants) | 101 | 100 | 97
units on a scale | -15.97 (1.313) | -13.03 (1.332) | -13.92 (1.354)
Statistical Analysis 1: Comparison: AZD6765 50 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.630, Mixed models for repeated measures — [p-value comment as in outcome 1, analysis 1]; LS mean difference = -2.05, 95% CI 2-sided [-5.628 to 1.522], Standard Error of Mean 1.816
Statistical Analysis 2: Comparison: AZD6765 100 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.630, Mixed models for repeated measures — [p-value comment as in outcome 1, analysis 1]; LS mean difference = 0.88, 95% CI 2-sided [-2.720 to 4.485], Standard Error of Mean 1.830

3. Secondary Outcome: Percentage of Patients With Sustained Response From Week 6 to Week 12 (Defined as ≥50% Reduction From Baseline in the MADRS Total Score at Week 6 and Which is Maintained Through Week 12)
Description: The percentage of patients with with Sustained Response (defined as ≥50% reduction from baseline in the MADRS total score at Week 6 and which is maintained through Week 12) was calculated.
Time Frame: Week 6 to Week 12
Population: The mITT analysis set included all randomized patients, who took IP and who have a non-missing baseline MADRS total score and at least 1 post-baseline MADRS total score, classified according to their randomized treatment.
Measure: Number; unit: percentage of participants analyzed
Arm/Group | AZD6765 50 mg | AZD6765 100 mg | Placebo
Number analyzed (Participants) | 101 | 100 | 97
percentage of participants analyzed | 22.8 | 23.0 | 21.6
Statistical Analysis 1: Comparison: AZD6765 50 mg vs Placebo; Logistic regression model including treatment as a fixed effect and the baseline MADRS total score as a covariate; Test type: Superiority or Other; p = 0.852, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.544 to 2.089], Standard Error of Mean 0.366
Statistical Analysis 2: Comparison: AZD6765 100 mg vs Placebo; Logistic regression model including treatment as a fixed effect and the baseline MADRS total score as a covariate; Test type: Superiority or Other; p = 0.821, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.552 to 2.115], Standard Error of Mean 0.370

4. Secondary Outcome: Percentage of Patients Who Were Responders (Defined as a ≥50% Reduction From Baseline in MADRS Total Score) at Week 6
Description: The percentage of patients who were Responders (defined as ≥50% reduction from baseline in MADRS total score) was calculated.
Time Frame: Baseline to Week 6
Population: as for outcome 3
Measure: Number; unit: percentage of participants analyzed
Arm/Group | AZD6765 50 mg | AZD6765 100 mg | Placebo
Number analyzed (Participants) | 86 | 84 | 82
percentage of participants analyzed | 36.0 | 44.0 | 39.0
Statistical Analysis 1: Comparison: AZD6765 50 mg vs Placebo; Generalized linear model of the repeated measures (GEE) with logic link including treatment, visit, and treatment by visit interaction as fixed effects and the baseline MADRS total score as a covariate; Test type: Superiority or Other; p = 0.751, GEE for repeated measures; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.485 to 1.686], Standard Error of Mean 0.318
Statistical Analysis 2: Comparison: AZD6765 100 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.555, GEE for repeated measures; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.650 to 2.233], Standard Error of Mean 0.315

5. Secondary Outcome: Percentage of Patients Who Were Responders (Defined as a ≥50% Reduction From Baseline in MADRS Total Score) at Week 12
Description: as for outcome 4
Time Frame: Baseline to Week 12
Population: as for outcome 3
Measure: Number; unit: percentage of participants analyzed
Arm/Group | AZD6765 50 mg | AZD6765 100 mg | Placebo
Number analyzed (Participants) | 89 | 85 | 81
percentage of participants analyzed | 48.3 | 36.5 | 40.7
Statistical Analysis 1: Comparison: AZD6765 50 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.434, GEE for repeated measures; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.699 to 2.301], Standard Error of Mean 0.304
Statistical Analysis 2: Comparison: AZD6765 100 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.286, GEE for repeated measures; Odds Ratio (OR) = 0.71, 95% CI 2-sided [0.377 to 1.334], Standard Error of Mean 0.322

6. Secondary Outcome: Percentage of Patients Who Were Remitted (Defined as MADRS Total Score ≤10) at Week 6
Description: The percentage of patients who were Remitted (defined as MADRS total score ≤10) was calculated.
Time Frame: Baseline to Week 6
Population: as for outcome 3
Measure: Number; unit: percentage of participants analyzed
Arm/Group | AZD6765 50 mg | AZD6765 100 mg | Placebo
Number analyzed (Participants) | 86 | 84 | 82
percentage of participants analyzed | 23.3 | 23.8 | 18.3
Statistical Analysis 1: Comparison: AZD6765 50 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.357, GEE for repeated measures; Odds Ratio (OR) = 1.42, 95% CI 2-sided [0.672 to 3.007], Standard Error of Mean 0.382
Statistical Analysis 2: Comparison: AZD6765 100 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.463, GEE for repeated measures; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.622 to 2.840], Standard Error of Mean 0.387

7. Secondary Outcome: Percentage of Patients Who Were Remitted (Defined as MADRS Total Score ≤10) at Week 12
Description: The percentage of patients who were Remitted (defined as MADRS total score ≤10) was calculated.
Time Frame: Baseline to Week 12
Population: as for outcome 3
Measure: Number; unit: percentage of participants analyzed
Arm/Group | AZD6765 50 mg | AZD6765 100 mg | Placebo
Number analyzed (Participants) | 89 | 85 | 81
percentage of participants analyzed | 27.0 | 22.4 | 25.9
Statistical Analysis 1: Comparison: AZD6765 50 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.911, GEE for repeated measures; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.532 to 2.031], Standard Error of Mean 0.342
Statistical Analysis 2: Comparison: AZD6765 100 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.509, GEE for repeated measures; Odds Ratio (OR) = 0.78, 95% CI 2-sided [0.382 to 1.613], Standard Error of Mean 0.368

8. Secondary Outcome: Change From Baseline in Functional Impairment as Measured by the Change From Baseline in the Sheehan Disability Scale (SDS) Total Score
Description: A 3-item, self-administered scale that measures the extent a patient is impaired by their disease. Higher scores indicate more severe impairment. The SDS total score is calculated as the sum of the score for the 3 intercorrelated domains (school/work, social life, and family life/home responsibilities), ranges from 0 (no impairment) to 30 (most severe impairment).
Time Frame: Baseline to Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | AZD6765 50 mg | AZD6765 100 mg | Placebo
Number analyzed (Participants) | 101 | 100 | 97
units on a scale
  Week 6 | -7.08 (0.959) | -6.90 (0.981) | -6.91 (0.989)
  Week 12 | -6.98 (0.995) | -6.80 (1.021) | -8.09 (1.034)
Statistical Analysis 1: Comparison: AZD6765 50 mg vs Placebo; MMRM includes treatment, pooled center, visit, treatment by visit interaction, and baseline SDS score by visit interaction as explanatory variables. Treatment, visit, treatment by visit interaction, and baseline SDS score by visit interaction are fixed effects in the model; pooled center is a random effect; Test type: Superiority or Other; p = 0.889, Mixed models for repeated measures — Analysis for change in SDS total score from baseline to Week 6; LS mean difference = -0.17, 95% CI 2-sided [-2.609 to 2.264], Standard Error of Mean 1.238
Statistical Analysis 2: Comparison: AZD6765 100 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.992, Mixed models for repeated measures — Analysis for change in SDS total score from baseline to Week 6; LS mean difference = 0.01, 95% CI 2-sided [-2.477 to 2.501], Standard Error of Mean 1.264
Statistical Analysis 3: Comparison: AZD6765 50 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.392, Mixed models for repeated measures — Analysis for change in SDS total score from baseline to Week 12; LS mean difference = 1.11, 95% CI 2-sided [-1.448 to 3.678], Standard Error of Mean 1.301
Statistical Analysis 4: Comparison: AZD6765 100 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.333, Mixed models for repeated measures — Analysis for changed in SDS total score from baseline to Week 12; LS mean difference = 1.29, 95% CI 2-sided [-1.327 to 3.908], Standard Error of Mean 1.329

9. Secondary Outcome: Change in Severity of Depressive Symptoms as Measured by Change From Baseline in the Clinical Global Impression-Severity (CGI-S) Score
Description: Clinical Global Impression - Severity (CGI-S) scale rates the severity of the patient's illness at the time of assessment, range from 1 (normal, not ill) to 7 (very severely ill).
Time Frame: Baseline to Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | AZD6765 50 mg | AZD6765 100 mg | Placebo
Number analyzed (Participants) | 101 | 100 | 97
units on a scale
  Week 6 | -1.5 (0.16) | -1.5 (0.16) | -1.4 (0.16)
  Week 12 | -1.8 (0.16) | -1.5 (0.16) | -1.6 (0.16)
Statistical Analysis 1: Comparison: AZD6765 50 mg vs Placebo; MMRM includes treatment, pooled center, visit, treatment by visit interaction, and baseline CGI-S score by visit interaction as explanatory variables. Treatment, visit, treatment by visit interaction, and baseline CGI-S score by visit interaction are fixed effects in the model; pooled center is a random effect; Test type: Superiority or Other; p = 0.728, Mixed models for repeated measures — Analysis for change in CGI-S total score from baseline to Week 6; LS mean difference = -0.1, 95% CI 2-sided [-0.49 to 0.34], Standard Error of Mean 0.21
Statistical Analysis 2: Comparison: AZD6765 100 mg vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.562, Mixed models for repeated measures — Analysis for change in CGI-S total score from baseline to Week 6; LS mean difference = -0.1, 95% CI 2-sided [-0.54 to 0.29], Standard Error of Mean 0.21
Statistical Analysis 3: Comparison: AZD6765 50 mg vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.283, Mixed models for repeated measures — Analysis for change in CGI-S total score from baseline to Week 12; LS mean difference = -0.2, 95% CI 2-sided [-0.64 to 0.19], Standard Error of Mean 0.21
Statistical Analysis 4: Comparison: AZD6765 100 mg vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.540, Mixed models for repeated measures — Analysis for changed in CGI-S total score from baseline to Week 12; LS mean difference = 0.1, 95% CI 2-sided [-0.29 to 0.55], Standard Error of Mean 0.21

10. Secondary Outcome: Change in Severity of Depressive Symptoms as Measured by the CGI-I Response (Defined as CGI-I Rating of "Very Much Improved" or "Much Improved") at Week 6
Description: A 3-part, clinician-administered scale that rates the improvement or worsening of the patient's illness from randomization (baseline). Each item is scored on a 1 to 7 scale. CGI-I scores >4 indicate worsening, while scores <4 indicate improvement.
Time Frame: Baseline to Week 6
Population: as for outcome 3
Measure: Number; unit: percentage of participants analyzed
Arm/Group | AZD6765 50 mg | AZD6765 100 mg | Placebo
Number analyzed (Participants) | 86 | 84 | 82
percentage of participants analyzed | 51.2 | 47.6 | 37.8
Statistical Analysis 1: Comparison: AZD6765 50 mg vs Placebo; Generalized linear model of the repeated measures (GEE) with logic link including treatment, visit, and treatment by visit interaction as fixed effects and the baseline CGI-S total score as a covariate; Test type: Superiority or Other; p = 0.067, GEE for repeated measures; Odds Ratio (OR) = 1.74, 95% CI 2-sided [0.962 to 3.141], Standard Error of Mean 0.302
Statistical Analysis 2: Comparison: AZD6765 100 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.230, GEE for repeated measures; Odds Ratio (OR) = 1.43, 95% CI 2-sided [0.798 to 2.558], Standard Error of Mean 0.297

11. Secondary Outcome: Change in Severity of Depressive Symptoms as Measured by the CGI-I Response (Defined as CGI-I Rating of "Very Much Improved" or "Much Improved") at Week 12
Description: as for outcome 10
Time Frame: Baseline to Week 12
Population: as for outcome 3
Measure: Number; unit: percentage of participants analyzed
Arm/Group | AZD6765 50 mg | AZD6765 100 mg | Placebo
Number analyzed (Participants) | 89 | 85 | 81
percentage of participants analyzed | 50.6 | 44.7 | 40.7
Statistical Analysis 1: Comparison: AZD6765 50 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.268, GEE for repeated measures; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.780 to 2.447], Standard Error of Mean 0.292
Statistical Analysis 2: Comparison: AZD6765 100 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.909, GEE for repeated measures; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.533 to 1.750], Standard Error of Mean 0.303

12. Secondary Outcome: Change From Baseline in Self-rated Severity of Depressive Symptoms as Measured by Quick Inventory of Depressive Symptomatology Self-Rated 16-item Scale (QIDS-SR-16) Total Score
Description: A 16-question self-report inventory that includes the 9 Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR) criteria symptom domains: sad mood, concentration, self-outlook, suicidal ideation, involvement, energy/fatigability, sleep disturbance (4 items: initial, middle, late insomnia, and hypersomnia), appetite/weight increased or decrease (4 items), and psychomotor agitation/retardation (2 items). The QIDS-SR-16 total scores range from 0 (least severe) to 27 (most severe).
Time Frame: Baseline to Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | AZD6765 50 mg | AZD6765 100 mg | Placebo
Number analyzed (Participants) | 101 | 100 | 97
units on a scale
  Week 6 | -8.7 (0.69) | -7.9 (0.70) | -8.1 (0.71)
  Week 12 | -9.2 (0.70) | -7.6 (0.71) | -8.9 (0.72)
Statistical Analysis 1: Comparison: AZD6765 50 mg vs Placebo; MMRM includes treatment, pooled center, visit, treatment by visit interaction, and baseline QIDS-SR-16 total score by visit interaction as explanatory variables. Treatment, visit, treatment by visit interaction, and baseline QIDS-SR-16 total score by visit interaction are fixed effects in the model; pooled center is a random effect; Test type: Superiority or Other; p = 0.505, Mixed models for repeated measures — Analysis for change in QIDS-SR-16 total score from baseline to Week 6; LS mean difference = -0.6, 95% CI 2-sided [-2.29 to 1.13], Standard Error of Mean 0.87
Statistical Analysis 2: Comparison: AZD6765 100 mg vs Placebo; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.842, Mixed models for repeated measures — Analysis for change in QIDS-SR-16 total score from baseline to Week 6; LS mean difference = 0.2, 95% CI 2-sided [-1.56 to 1.91], Standard Error of Mean 0.88
Statistical Analysis 3: Comparison: AZD6765 50 mg vs Placebo; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.788, Mixed models for repeated measures — Analysis for change in QIDS-SR-16 total score from baseline to Week 12; LS mean difference = -0.2, 95% CI 2-sided [-1.98 to 1.51], Standard Error of Mean 0.89
Statistical Analysis 4: Comparison: AZD6765 100 mg vs Placebo; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.133, Mixed models for repeated measures — Analysis for changed in QIDS-SR-16 total score from baseline to Week 12; LS mean difference = 1.4, 95% CI 2-sided [-0.42 to 3.12], Standard Error of Mean 0.90

ADVERSE EVENTS:
Description: The AZD6765iv (intravenous) 100 mg group had one less subject than the numbers provided in the Participant Flow Module because one subject who was randomized did not receive any study medication and thus was excluded from the efficacy and safety analysis sets.
Groups:
- AZD6765iv 100 mg; AZD6765iv 50 mg; Placebo: Intravenous infusion
Arm/Group | AZD6765iv 100 mg | AZD6765iv 50 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 4/100 | 2/101 | 4/100
Other Adverse Events (participants affected / at risk) | 68/100 | 59/101 | 47/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD6765iv 100 mg (N=100) | AZD6765iv 50 mg (N=101) | Placebo (N=100)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1)
HEPATITIS C (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
DEPRESSIVE SYMPTOM (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
INTENTIONAL DRUG MISUSE (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
MAJOR DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
SUICIDE ATTEMPT (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD6765iv 100 mg (N=100) | AZD6765iv 50 mg (N=101) | Placebo (N=100)
CONSTIPATION (Gastrointestinal disorders) | 6 (6) | 2 (2) | 5 (5)
DIARRHOEA (Gastrointestinal disorders) | 5 (7) | 7 (10) | 5 (6)
DRY MOUTH (Gastrointestinal disorders) | 6 (17) | 3 (5) | 2 (3)
NAUSEA (Gastrointestinal disorders) | 21 (26) | 13 (13) | 13 (16)
FATIGUE (General disorders) | 6 (6) | 5 (6) | 5 (6)
FEELING DRUNK (General disorders) | 6 (38) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 6 (7) | 7 (8) | 4 (4)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 7 (9) | 2 (2)
DIZZINESS (Nervous system disorders) | 45 (205) | 27 (63) | 10 (17)
HEADACHE (Nervous system disorders) | 17 (29) | 20 (28) | 18 (28)
SEDATION (Nervous system disorders) | 7 (26) | 5 (18) | 5 (13)
SOMNOLENCE (Nervous system disorders) | 6 (12) | 9 (16) | 7 (9)
DISSOCIATION (Psychiatric disorders) | 8 (37) | 4 (6) | 4 (7)
INSOMNIA (Psychiatric disorders) | 6 (6) | 5 (6) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less